CLINICAL TRIAL: NCT00447811
Title: Two Ascending Single Doses Crossover, Placebo Controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MOA-728 Administered Orally to Subjects on Stable Methadone Maintenance
Brief Title: Study Evaluating MOA-728 in Subjects on Stable Methadone Maintenance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3200A3-1109
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Methadone-maintenance Subjects
Keywords: Methadone

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
This is a study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of MOA-728 in subjects on stable methadone maintenance.

ELIGIBILITY:
Inclusion Criteria:

* History of methadone treatment for at least 1 month before day -1 at a dose of ≥ 30 mg/day, and a positive drug test result for methadone.
* Healthy as determined by the investigator on the basis of screening evaluations.

Exclusion Criteria:

* Allergy to opioids (eg, codeine, morphine, or oxymorphone) or opioid antagonists (eg, naloxone or naltrexone).
* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics

SECONDARY OUTCOMES:
Safety, tolerability, and pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Willingboro, New Jersey, United States